CLINICAL TRIAL: NCT06174974
Title: The Effect of Education Given to Patients Before Cardiac Surgery on Environmental Stressors Perceived by the Patient: A Randomised Controlled Study
Brief Title: The Effect of Education on Environmental Stressors Perceived by Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeynep Kızılcık Ozkan, Assistant professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/297
Record Dates: First submitted 2023-11-27; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Education Of Patients
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The patients in the experimental group will be informed by the researcher in the training room in the ward 1 day before the operation (verbal permission was obtained) with an educational presentation on intensive care unit stressors.
  Patients in the control group will not be given preoperative training on intensive care unit stressors by the researcher. Patients in the control group will receive standard care*.
Who Masked: Outcomes Assessor
Masking Description: The data will be collected and coded by the nurse researcher. Data will be analyzed by an independent statistician. The study groups will be disguised as A and B. The statistician will not know the groups. In addition, the statistical expert will not see the data of the experimental group regarding satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients in the experimental group will be informed by the researcher in the training room in the ward 1 day before the operation (verbal permission was obtained) with an educational presentation on intensive care unit stressors.
  Interventions: Other: Education
- Control group (No Intervention): Patients in the control group will not be given preoperative training on intensive care unit stressors by the researcher. Patients in the control group will receive standard care*.

INTERVENTIONS:
Other: Education — The education was designed to cover the environmental stressors of the intensive care unit and the practices performed to reduce these stressors. The education content was created according to the Activities of Daily Living (ADL) Theory based on the institution's cardiovascular surgical intensive care unit protocols (Cardiovascular surgical intensive care unit visitor entry-exit rules information form) and the literature (included at the end of the presentation). Expert (intensive care nurses, ward nurses, cardiovascular surgeons and academic nurses) opinions were obtained. Patient-friendly and simple language was used to ensure that the content of the information presentation was acceptable and interesting.
  Arms: Experimental group

SUMMARY:
Aim of the Thesis and Hypotheses: (The aim of the thesis and hypotheses should be stated in detail.) In this study, it was aimed to determine the effect of the education given to the patients before cardiac surgery on the environmental stressors perceived by the patients in the intensive care unit.

H1: The education given before heart surgery has an effect on the environmental stressors perceived by patients in the intensive care unit.

H2: The education given before cardiac surgery has no effect on the environmental stressors perceived by patients in the intensive care unit.

DETAILED DESCRIPTION:
The randomised controlled trial will be conducted in the cardiovascular surgery service of Trakya University Health Research and Application Centre. Date of research will be conducted: November.2023- March 2024 The research sample will consist of 64 volunteer patients. The sample was determined using power analysis at the research planning stage. The minimum number of people to be included in the sample was calculated as 54, each group consisting of 27 (1:1) patients, with an effect size of 0.80, 95% confidence level, 5% tolerance and 80% power ratio, using the G.Power 3.1.9.4 programme. In case of possible patient loss, the sample size was increased by 20% and each group was decided to consist of 32 patients. A total of 64 patients were included in the sample.

Data Collection Forms Patient information form; The form was developed by the researchers in line with the literature and includes some characteristics (age, gender, educational status, marital status, habits, surgical experience, presence of preoperative stress, physician diagnosis, surgical procedure performed, presence of chronic disease, presence of companion, presence of intensive care experience, perception of intensive care experience, opinion about the concept of intensive care, presence of anxiety about intensive care follow-up, postoperative hospitalisation day in the intensive care unit).

Intensive Care Unit Environmental Stressors Scale; This scale was developed by Ballard (1) in 1981 to describe the stressors perceived by patients treated in intensive care units and revised by Cochran and Ganong (2) in 1989. The scale was adapted into Turkish by Çınar, Aslan and Kurtoğlu (3) and Cronbach's alpha value was found to be 0.94. The scale contains 42 items and the answers are in 4-point Likert type. 1=Never affects, 2= Very little affects, 3= Frequently affects, 4= Very much affects. The lowest total score of the scale is 42 points and the highest is 168 points.

Patient satisfaction form; The satisfaction of the patients in the experimental group with the preoperative training will be evaluated with a numerical rating scale ranging from 0 to 10 points (0 = Not at all satisfied, 10 = Very satisfied).

Data Collection Process The researcher will visit the service and identify the patients who will undergo cardiac surgery. Before starting data collection, the eligibility of the patients will be determined based on the sampling criteria. Patients who meet the inclusion criteria will be informed verbally and in writing about the research, scales, etc. in the preoperative period and the informed consent form will be signed. "Patient Information Form" will be applied in the preoperative period. The data of the study will be collected by the researcher in the patient room by face-to-face interview method.

Patients in the control group will not be given preoperative training on intensive care unit stressors by the researcher. Patients in the control group will receive standard care. Patients transferred from the cardiovascular surgery intensive care unit to the cardiovascular surgery service after surgery will be visited by the researcher on the day of transfer and the appropriate time for data collection will be determined by appointment between the patient and the researcher. The researcher will come to the cardiovascular surgery service again at the appointment time and apply the "Intensive Care Unit Environmental Stressors Scale".

Patients in the experimental group will be informed by the researcher in the training room in the ward 1 day before the surgery (verbal permission was obtained) with a training presentation on intensive care unit stressors.Patients transferred from the cardiovascular surgery intensive care unit to the cardiovascular surgery service after surgery will be visited by the researcher on the day of transfer and the "Intensive Care Unit Environmental Stressors Scale" will be applied. In addition, patients' satisfaction with the preoperative education will be evaluated.

The training lasts approximately 15-20 minutes.The training will be presented by transferring to the television screen in the room via flash memory. The training will be presented by transferring to the television screen in the patient education room via flash memory. While the researcher verbally conveys the information on the slides to the patients and their relatives, the education will be strengthened by ensuring that the patients follow the slides enriched with visual content.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment in the cardiovascular surgery ward prior to surgery,
* Undergoing planned cardiac surgery under general anaesthesia,
* Admitted to the cardiovascular surgery intensive care unit after surgery,
* At least 24 hours in the intensive care unit,
* Sternotomy performed,
* who volunteered to participate in the research,
* No mental disability,
* 18 years of age,
* Literate,
* Accepting random selection,
* Patients without communication problems in Turkish

Exclusion Criteria:

* Treated as a day patient in the cardiovascular surgery ward,
* Pre-operative inpatient treatment in cardiology, coronary intensive care or other external wards,
* Without sternotomy,
* Admitted to intensive care or external ward after surgery,
* Emergency surgery,
* Not volunteering to participate in the research,
* Mentally handicapped,
* Under 18 years of age,
* Illiterate,
* which does not accept random selection,
* Patients with communication problems in Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
environmental stressors perceived by patients | Patients transferred from the cardiovascular surgery intensive care unit to the cardiovascular surgery service, on the day of transfer (postoperative 2-3rd day).
  To determine the effect of education given before cardiac surgery on environmental stressors perceived by patients in the intensive care unit."Intensive Care Unit Environmental Stressors Scale" will be applied on the day the patients are transferred to the ward. The 4-Likert type scale consists of 42 items. The items evaluated as "It does not affect at all (1 point) ", "It affects very little (2 points)", "It frequently affects (3 points)" and "It affects too much (4 points)". The lowest total score is 42 and the highest total score is 168. The high score obtained from the scale indicates that there are many environmental stressors in the intensive care environment, and they negatively affect the patients.

SECONDARY OUTCOMES:
patients' satisfaction | postoperative period (postoperative 2nd or 3rd day)
  To determine the effect of education given before cardiac surgery on patients' satisfaction. Patient satisfaction form; The satisfaction of the patients in the experimental group with the preoperative training will be evaluated with a numerical rating scale ranging from 0 to 10 points (0 = Not at all satisfied, 10 = Very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Trakya University, Edirne, Turkey (Türkiye)